CLINICAL TRIAL: NCT00815503
Title: Postoperative Analgesia With Local Infiltration After Periacetabular Osteotomy For The Treatment Of Dysplasia
Brief Title: Postoperative Analgesia With Local Infiltration After Periacetabular Osteotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Rune Bech, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S20080152
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Periacetabular Osteotomy; Pain
Keywords: Anesthetics; Local infiltration; Periacetabular osteotomy
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine
- Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine — Approved by the Danish Medicines Agency
  Arms: Ropivacaine
Drug: Placebo — Saline
  Arms: Saline

SUMMARY:
Pain treatment after periacetabular osteotomy is traditionally based on systemic opioids wich have side effects. The purpose of this study is to evaluate the analgetic effect of wound infiltration with local anaesthesia after periacetabular osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Periacetabular osteotomy due to traditional dysplasia or retroverted acetabulum
* Informed consent

Exclusion Criteria:

* Intolerance of local anaesthesia
* Habitual use of opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Consumption of rescue analgetics | Assesment of opioid rescue analgetics every 24 hours for 14 days postoperatively

SECONDARY OUTCOMES:
Pain | Assessment of pain four times every day for five days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Bech RD, Ovesen O, Lindholm P, Overgaard S. Local anesthetic wound infiltration for pain management after periacetabular osteotomy. A randomized, placebo-controlled, double-blind clinical trial with 53 patients. Acta Orthop. 2014 Apr;85(2):141-6. doi: 10.3109/17453674.2014.899840. PMID 24650022